CLINICAL TRIAL: NCT02605551
Title: The Utilization of Osteopathic Manipulation (OMT) as an Adjunct Therapy in the Treatment of Hypertension
Brief Title: Hypertension and Osteopathic Treatment
Acronym: HOT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Period Ended / Not Completed
Sponsor: Larkin Community Hospital (Other)
Collaborators: Miami Beach Community Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCH-2-022015
Record Dates: First submitted 2015-11-07; First posted 2015-11-16 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Prehypertension; Hypertension; Osteopathic Manipulation; Sympathetic Nervous System
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMT Group (Active Comparator): During the initial visit, the subject will have his BP recorded manually by the osteopathic physician in a standardized fashion. The subject will then undergo the OMT protocol and have his BP recorded again immediately afterwards. This will represent the conclusion of the initial visit. There will be 2 subsequent visits about 2-3 weeks apart that will be identical to this visit. Following the third visit, the next follow-up will be 2 months afterwards. However, the patient will only have his BP checked, and will not undergo an OMT treatment. The final visit will be another 2 months afterwards and will also be a simple BP check with no OMT treatment. The principles of lifestyle modification (diet/exercise/weight loss) will also be discussed at each visit.
  Interventions: Procedure: Osteopathic Manipulative Therapy; Behavioral: Lifestyle Modification
- Control Group (Placebo Comparator): Patients in this arm will only receive lifestyle modification recommendations at each visit, along with a BP check. No antihypertensive medication changes will be made unless indicated by the guidelines.
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Procedure: Osteopathic Manipulative Therapy — All OMT techniques will be performed by osteopathic physicians who will have received training specific to this protocol prior to study initiation. All used techniques will be slow moving and gentle to augment rest and relaxation, promote autonomic balance, and release fascial contractures. The techniques that will be used in this protocol are:
  1. OM Occipitomastoid release technique
  2. Sub-Occipital Release Technique
  3. Rib Raising Technique
  4. Rotatory stimulation of posterior Chapman's Reflexes
  5. Lymphatic Pumps and Effleurage: (Pedal Pump of Dalrymple)
  Other Names: OMT; OMM; NMM; Osteopathic Manipulation Treatment; Osteopathic Manipulation Medicine; Neuromusculoskeletal Medicine; Neuromuscular Medicine
  Arms: OMT Group
Behavioral: Lifestyle Modification — Patients will be counseled on healthy behaviors such as regular exercise, weight loss, and a healthy diet

SUMMARY:
The goal of this study is to demonstrate the use of osteopathic manipulative therapy (OMT) in the effective management of hypertension. The investigators hypothesize that by addressing/correcting somatic dysfunctions with OMT, the sympathetic overdrive that could be the root cause of the elevation in blood pressure will be downregulated. If this is the case, then an effective therapy for hypertension could indeed be regular OMT treatment. This could also result in the avoidance of potentially harmful antihypertensive medications which comprise a majority of the current therapeutic strategy in the treatment of hypertension (along with lifestyle modification). A third implication of the results of this project could be a reduction in the progression of this disease. Under the current standard of care, a majority of hypertensive patients only experience a worsening of the disease over time under the current therapeutic guidelines.

DETAILED DESCRIPTION:
Approximately 60% of American adult population has prehypertension or hypertension. Subgroups such as African Americans, elderly, low-socioeconomic-status, and the overweight population, are disproportionately affected. Larkin Community Hospital (LCH) and its affiliated sites provide a great number of patients in these particular subgroups and this represents an ideal institution to study this tremendous health issue. Hypertension is a progressive disease and it has been shown·that, later in life, patients with borderline hypertension will progress at a much higher rate to Stage 1 or 2 hypertension as compared with normotensive population. The Framingham study has been demonstrated after 26 years of follow up, that 71% of patients with high-normal blood pressure (systolic, 130-139 mm Hg; diastolic, 85-89) developed clinical hypertension later in life. The Tecumseh blood pressure study has shown that subjects aged between 20 and 40 years old with borderline hypertension (average BP 130.7/93.8) have had significantly higher childhood (average age 6 years) BP levels compared with normotensive ones, further illustrating the propensity of this disease to progress. Also, the bell-shaped curve of blood pressure in the general population shows that the largest group of people will have blood pressures in the prehypertensive range, showing what a large proportion of the population would be affected by advances in the management of this disease.

Osteopathic manipulative therapy (OMT) is a therapeutic modality utilized by osteopathic physicians to address somatic dysfunctions in the musculoskeletal system. Somatic dysfunctions are abnormalities in musculoskeletal tissue texture and intervertebral joint dysfunction. Close associations between spinal vertebrae and the autonomic nervous system via the sympathetic trunk and ganglia are believed to be one of the mechanisms by which musculoskeletal system changes can affect other organs (somatovisceral reflex). Indeed, osteopathic philosophy posits that OMT has a distinct effect beyond the musculoskeletal system. Additionally, the autonomic and lymphatic systems and their effects upon the function of the cardiovascular system have been extensively studied. OMT has been shown by Stiles to significantly decrease both mortality and morbidity of patients with cardiovascular dysfunctions. Rogers et al. have also reported that OMT has been demonstrated to be of significant value in some patients with coronary insufficiency.

The bulk of the sympathetic nervous system lies adjacent to the thoracic spine as well as the superior lumbar spine. Particularly, the sympathetic innervation of the heart has its origins in cord segments T1-T6, with synapses occurring between pre-and post-ganglionic fibers in the upper thoracic and/or cervical ganglia. As previously discussed, alterations in the spinal mechanics and the presence of somatic dysfunctions in these regions of the spine have been theorized to alter the function of the autonomic nervous system originating from these regions. Specific cardiovascular effects of these dysfunctions are increased heart rate, increased contractility, increased cardiac work-load, and increased total peripheral resistance. To provide further evidence of the link between the musculoskeletal system and the cardiovascular system, it was demonstrated that patients with Travell triggerpoints in the right pectoralis muscle may be prone to periods of supraventricular tachyarrhythmias. When these trigger points are the etiologies of the arrhythmias, the arrhythmia disappears when the trigger point is effectively treated.

The goal of this study is to demonstrate the use of OMT in the effective management of hypertension. The investigators hypothesize that by addressing/correcting somatic dysfunctions with OMT, it will downregulate the sympathetic overdrive that could be the root cause of the elevation in blood pressure. If this is the case, then an effective therapy for hypertension could indeed be regular OMT treatment. This could also result in the avoidance of potentially harmful antihypertensive medications which comprise a majority of the current therapeutic strategy in the treatment of hypertension (along with lifestyle modification). A third implication of the results of this project could be a reduction in the progression of this disease. As discussed above, a majority of hypertensive patients only experience a worsening of the disease over time under the current therapeutic guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure meeting the criteria for pre-hypertension (130-139/85-89) or stage 1 hypertension (140-159/90-99) at two different instances
* Otherwise healthy adult patients consenting to study participation

Exclusion Criteria:

* Presence of co-morbid renal or liver disease
* medication regimen of more than one anti-hypertensive medication
* Presence of pre-existing heart disease, CAD (coronary artery disease), severe stenotic valvular disease, CHF (congestive heart failure), cardiomyopathy
* Presence of condition that would make application of OMT protocol impossible
* Pregnancy
* Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-01 (Estimated); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 14 weeks
  Participants will have an initial BP measurement, followed by measurements at 2, 4 and 6 weeks (both before and after OMT treatment performed at those visits). Then, they will have a simple BP check at 10 weeks and finally at 14 weeks. The goal of these measurements is to ascertain whether or not there is a change of baseline systolic/diastolic BP with serial OMT treatments

CONTACTS AND LOCATIONS:
Overall Officials: Rohit S Mehra, DO, MPH, MS, Principal Investigator — Larkin Community Hospital; David Stuckey, DO, Study Director — Larkin Community Hospital; Scott E Spagnolo-Hye, DO, MS, Study Chair — Larkin Community Hospital

REFERENCES:
- [Background] Daiber WF: Disorders of the Kidneys in Hoag JM (ed) Osteopathic Medicine. New York, McGraw-Hill, 1969, Ch 39, PP644-5
- [Background] Wang Y, Wang QJ. The prevalence of prehypertension and hypertension among US adults according to the new joint national committee guidelines: new challenges of the old problem. Arch Intern Med. 2004 Oct 25;164(19):2126-34. doi: 10.1001/archinte.164.19.2126. PMID 15505126
- [Background] Julius S, Schork MA. Borderline hypertension--a critical review. J Chronic Dis. 1971 Mar;23(10):723-54. doi: 10.1016/0021-9681(71)90005-1. No abstract available. PMID 4933751
- [Background] Leitschuh M, Cupples LA, Kannel W, Gagnon D, Chobanian A. High-normal blood pressure progression to hypertension in the Framingham Heart Study. Hypertension. 1991 Jan;17(1):22-7. doi: 10.1161/01.hyp.17.1.22. PMID 1986979
- [Background] Julius S, Jamerson K, Mejia A, Krause L, Schork N, Jones K. The association of borderline hypertension with target organ changes and higher coronary risk. Tecumseh Blood Pressure study. JAMA. 1990 Jul 18;264(3):354-8. PMID 2362331
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] The Foundations of Osteopathic Medicine, 3rd edition. Lippincott, Williams, and Wilkins. 2010. ISBN 0781766710
- [Background] Fitzgerald M, Stiles, E: Osteopathic Hospitals' solution to DRGs may be OMT. The DO Nov. 1984: 97-101
- [Background] Rogers JT, Rogers JC. The role of osteopathic manipulative therapy in the treatment of coronary heart disease. J Am Osteopath Assoc. 1976 Sep;76(1):21-31. No abstract available. PMID 1048963
- [Background] Lown B, Verrier RL, Rabinowitz SH. Neural and psychologic mechanisms and the problem of sudden cardiac death. Am J Cardiol. 1977 May 26;39(6):890-902. doi: 10.1016/s0002-9149(77)80044-1. PMID 860697
- [Background] Cox JM, Gorbis S, Dick LM, Rogers JC, Rogers FJ. Palpable musculoskeletal findings in coronary artery disease: results of a double-blind study. J Am Osteopath Assoc. 1983 Jul;82(11):832-6. No abstract available. PMID 6885531